CLINICAL TRIAL: NCT00114738
Title: Randomized Phase II Study of Dose-Adjusted EPOCH-Rituximab-Bortezomib (EPOCH-R-B) Induction Followed by Bortezomib Maintenance Versus Observation in Untreated Mantle Cell Lymphoma With Microarray Profiling and Proteomics
Brief Title: EPOCH-R Chemotherapy Plus Bortezomib to Treat Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wyndham Wilson, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 050170; 05-C-0170; NCT00131976 (obsolete NCT alias)
Record Dates: First submitted 2005-06-17; First posted 2005-06-17 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Lymphoma, Mantle Cell; Mantle Cell Lymphoma
Keywords: Proteasome Inhibition; NF-Kappa-B; Gene Expression Signature; Cyclin D1; Translational Studies; Lymphoma; Mantle Cell Lymphoma; MCL
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — Rituximab; Bortezomib; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- EPOCH-R + Bortezomib (Experimental): Combo chemo etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH)-Rituxan (R) + Bortezomib (B)
  Interventions: Drug: Rituximab (R); Biological: EPOCH; Drug: Bortezomib
- Bortezomib "window" (Experimental): Bortezomib alone
  Interventions: Drug: Bortezomib (B)
- Bortezomib maintenance (Active Comparator): Bortezomib maintenance
  Interventions: Drug: Bortezomib
- Observation (Other): At the beginning of part C patients are randomized to receive bortezomib maintenance or observation without bortezomib.
  Interventions: Drug: Bortezomib or observation

INTERVENTIONS:
Drug: Rituximab (R) — Rituximab is given with etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) and bortezomib every 3 weeks for 6 cycles.
  Other Names: Rituxan
  Arms: EPOCH-R + Bortezomib
Biological: EPOCH — EPOCH is given with Rituximab and bortezomib every 3 weeks for 6 cycles.
  Arms: EPOCH-R + Bortezomib
Drug: Bortezomib (B) — Bortezomib is given alone for one cycle.
  Other Names: Velcade
  Arms: Bortezomib "window"
Drug: Bortezomib — Bortezomib is given with EPOCH and rituximab every 6 weeks for 12 cycles.
  Other Names: Velcade
  Arms: Bortezomib maintenance; EPOCH-R + Bortezomib
Drug: Bortezomib or observation — At the beginning of Part C, patients are randomized to receive bortezomib maintenance or be observed w/o bortezomib.
  Other Names: Velcade
  Arms: Observation

SUMMARY:
This study will evaluate the effectiveness of etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin-rituximab (EPOCH-R) chemotherapy plus bortezomib for treating mantle cell lymphoma, a cancer of white blood cells called lymphocytes. EPOCH-R consists of the drugs prednisone, etoposide, doxorubicin and vincristine, with the addition of a new drug called rituximab. In a recent study of patients with newly diagnosed mantle cell lymphoma, 92 percent had a complete remission of their disease after treatment with EPOCH-R. This study will test whether adding bortezomib as "maintenance therapy" once chemotherapy is finished will lengthen the time before the disease relapses and improve the overall cure rate.

Patients 18 years of age and older with mantle cell lymphoma may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, electrocardiogram, multi-gated acquisition scan (MUGA) or echocardiogram, imaging studies and biopsy to determine the extent of disease, and possible colonoscopy.

Participants undergo treatment in three parts, as follows:

* Part 1: Bortezomib alone: Patients receive 4 doses of bortezomib over 3 weeks. The drug is injected into a vein over about 30 seconds.
* Part 2: EPOCH-R chemotherapy plus bortezomib: This phase of treatment begins 3 to 4 weeks after completing Part 1. Treatment is given on an outpatient basis in six 3-week cycles, with all drugs administered over the first 5 days of each cycle. Patients take prednisone by mouth on days 1 to 5 and etoposide, doxorubicin, and vincristine as a 96-hour infusion through a vein over days 1 to 5. The infused drugs are delivered through a lightweight, portable infusion pump. Rituximab is given by vein over several hours on day 1 immediately before the chemotherapy infusion begins. Bortezomib is given by vein over 30 seconds on day 1 before the rituximab and again on day 4. Cyclophosphamide is given by vein over about 15 minutes on day 5 immediately after the chemotherapy infusion is completed. Patients are taught how to self inject granulocyte colony stimulating factor (G-CSF), a drug that helps boost white cell counts after chemotherapy. They inject the drug under the skin (like an insulin shot) for 10 days of each cycle beginning day 6. Patients also take an antibiotic to help prevent infection during chemotherapy.
* Part 3: Bortezomib alone: After completing EPOCH-R-B therapy, patients are randomly assigned to receive or not to receive bortezomib alone. The drug is given in 2 doses over 5 days, with a break of 16 days before the next dose. These 3-week cycles continue for up to 18 months or until the disease comes back or worsens. Patients who are assigned to the group that does not receive bortezomib will be offered the drug if their disease relapses.

During therapy, patients have tests performed on their bone marrow, tumor tissue, blood or other fluids to look at different genes and proteins that may be involved in the development of their lymphoma or the reaction of the immune system. A tissue biopsy is done before treatment begins and a day after treatment starts. Disease progress is followed with computed tomography (CT) scans and blood tests. When treatment is completed, patients whose cancer has disappeared are scheduled for periodic follow-up examinations and tests. Those whose disease remains or recurs may be offered participation in another protocol if an appropriate one is available or are returned to the care of their local physician.

...

DETAILED DESCRIPTION:
Background:

Mantle cell lymphoma (MCL) presents a clinical challenge because it is aggressive and incurable with chemotherapy. Therefore novel treatment approaches are needed.

MCL has overexpression of NF-kappa B (NF-kappa B), a transcription factor that affects cell growth and survival, and cyclin D1 that affects cell cycle and growth. These proteins appear to be involved in the pathogenesis of MCL.

Bortezomib, a proteasome inhibitor that inhibits NF-kappa B and cyclin D1, has demonstrated activity in patients with relapsed or refractory MCL.

Dose-adjusted-etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin-rituximab (EPOCH-R) has excellent activity in MCL, with a complete response (CR) rate of 92%, but patients eventually relapse.

Objective:

Determine the progression free survival (PFS) and overall survival (OS) of dose-adjusted etoposide, doxorubicin, and cyclophosphamide with vincristine, prednisone, and rituximab,bortezomib (DA-EPOCH-RB) followed by bortezomib maintenance versus observation.

Eligibility:

Diagnosis of mantle cell lymphoma.

No prior treatment except for local radiation or a short course of steroids for control of symptoms,

Age greater than or equal to 18 years old.

Adequate major organ function unless impairment is due to lymphoma.

Study Design:

To assess the clinical activity and biological effects of bortezomib, patients will initially receive one cycle of bortezomib alone with sequential tumor biopsies for microarray analysis.

All patients will then receive Dose-adjusted (DA)-EPOCH-RB for 6 cycles, and if they have at least a PR, this will be followed by randomization to either immediate bortezomib maintenance x 18 months, or to observation, followed by bortezomib if progression occurs. This study has as a primary goal, to describe progression free survival (PFS) and overall survival of early bortezomib maintenance versus observation following induction with bortezomib followed by DA-EPOCH-RB. Important secondary goals are to assess response and toxicity to bortezomib alone or DA-EPOCH-RB, to evaluate time to progression after receiving bortezomib following progression on an observation arm, and to assess the biological effects of bortezomib on untreated MCL.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Diagnosis of mantle cell lymphoma (confirmed at National Cancer Institute (NCI)). All variants are eligible.

Age greater than or equal to 18 years.

No prior treatment except for local radiation or a short course of steroids for control of symptoms.

All stages of disease.

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 3.

Adequate major organ function (serum creatinine less than or equal to 1.5 mg/dl or creatinine clearance greater than 50 ml/min; bilirubin less than 2 mg/dl (total) except less than 5 mg/dl in patients with Gilbert's syndrome as defined by greater than 80% unconjugated; Absolute neutrophil count (ANC) greater than 1000 and platelets greater than 75,000) unless impairment due to organ involvement by lymphoma.

No myocardial infarction within 6 months prior to enrollment or New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiogram (ECG) abnormality at Screening has to be documented by the investigator as not medically relevant.

No grade 2 greater than or equal to peripheral neuropathy within 14 days before enrollment.

Ability to give informed consent.

Human immunodeficiency virus (HIV) antibody negative.

Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Female subject is not pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-human chorionic gonadotropin (hCG)) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women

Male subject agrees to use an acceptable method for contraception for the duration of the study.

No history of a prior invasive malignancy in past 5 years

No known involvement of central nervous system by lymphoma

No history of hypersensitivity to boron or mannitol.

Patient has not received other investigational drugs with 14 days before enrollment.

No serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Exclusion for fludeoxyglucose (FDG) scan is anyone exceeding the weight limit of the scanner (350 lb).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-06-15 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H Wilson, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Velders GA, Kluin-Nelemans JC, De Boer CJ, Hermans J, Noordijk EM, Schuuring E, Kramer MH, Van Deijk WA, Rahder JB, Kluin PM, Van Krieken JH. Mantle-cell lymphoma: a population-based clinical study. J Clin Oncol. 1996 Apr;14(4):1269-74. doi: 10.1200/JCO.1996.14.4.1269. PMID 8648383
- [Background] Campo E, Raffeld M, Jaffe ES. Mantle-cell lymphoma. Semin Hematol. 1999 Apr;36(2):115-27. PMID 10319380
- [Background] Hiddemann W, Unterhalt M, Herrmann R, Woltjen HH, Kreuser ED, Trumper L, Reuss-Borst M, Terhardt-Kasten E, Busch M, Neubauer A, Kaiser U, Hanrath RD, Middeke H, Helm G, Freund M, Stein H, Tiemann M, Parwaresch R. Mantle-cell lymphomas have more widespread disease and a slower response to chemotherapy compared with follicle-center lymphomas: results of a prospective comparative analysis of the German Low-Grade Lymphoma Study Group. J Clin Oncol. 1998 May;16(5):1922-30. doi: 10.1200/JCO.1998.16.5.1922. PMID 9586911
- [Derived] Lakhotia R, Melani C, Dunleavy K, Pittaluga S, Saba N, Lindenberg L, Mena E, Bergvall E, Lucas AN, Jacob A, Yusko E, Steinberg SM, Jaffe ES, Wiestner A, Wilson WH, Roschewski M. Circulating tumor DNA predicts therapeutic outcome in mantle cell lymphoma. Blood Adv. 2022 Apr 26;6(8):2667-2680. doi: 10.1182/bloodadvances.2021006397. PMID 35143622
- [Derived] Chang BY, Francesco M, De Rooij MF, Magadala P, Steggerda SM, Huang MM, Kuil A, Herman SE, Chang S, Pals ST, Wilson W, Wiestner A, Spaargaren M, Buggy JJ, Elias L. Egress of CD19(+)CD5(+) cells into peripheral blood following treatment with the Bruton tyrosine kinase inhibitor ibrutinib in mantle cell lymphoma patients. Blood. 2013 Oct 3;122(14):2412-24. doi: 10.1182/blood-2013-02-482125. Epub 2013 Aug 12. PMID 23940282
- [Derived] Perez-Galan P, Mora-Jensen H, Weniger MA, Shaffer AL 3rd, Rizzatti EG, Chapman CM, Mo CC, Stennett LS, Rader C, Liu P, Raghavachari N, Stetler-Stevenson M, Yuan C, Pittaluga S, Maric I, Dunleavy KM, Wilson WH, Staudt LM, Wiestner A. Bortezomib resistance in mantle cell lymphoma is associated with plasmacytic differentiation. Blood. 2011 Jan 13;117(2):542-52. doi: 10.1182/blood-2010-02-269514. Epub 2010 Oct 18. PMID 20956803
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-C-0170.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib Then Bortezomib + DA-EPOCH-R Induction: Bortezomib is given alone for one cycle, then combo chemo etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH)-Rituxan (R) + Bortezomib (B) is given every 3 weeks for 6 cycles.
- Bortezomib Maintenance: Bortezomib alone is given in 3 week cycles. 3-week cycles continue up to 18 months or until the disease comes back or worsens.
- Observation: Participants are observed without treatment.
Period: Bortezomib Then Bortezomib + Induction
Arm/Group | Bortezomib Then Bortezomib + DA-EPOCH-R Induction | Bortezomib Maintenance | Observation
Started | 53 | 0 | 0
Started With Bortezomib Alone | 47 | 0 | 0
Skipped Bortezomib Alone | 6 | 0 | 0
Completed | 51 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0
Period: Screening for Randomization
Arm/Group | Bortezomib Then Bortezomib + DA-EPOCH-R Induction | Bortezomib Maintenance | Observation
Started | 51 | 0 | 0
Completed | 30 | 0 | 0
Not Completed | 21 | 0 | 0
Not completed — Neuropathy | 17 | 0 | 0
Not completed — Progressive disease | 2 | 0 | 0
Not completed — CNS Hemorrhage | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Randomization
Arm/Group | Bortezomib Then Bortezomib + DA-EPOCH-R Induction | Bortezomib Maintenance | Observation
Started | 0 | 14 | 16
Completed | 0 | 14 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All Participants who received at least one dose of Bortezomib alone followed by EPOCH-R+B chemotherapy.
  Bortezomib (B): Bortezomib is given alone for one cycle.
  Combo chemo etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH)-Rituxan (R) + Bortezomib (B)
  Rituximab (R): Rituximab is given with etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) and bortezomib every 3 weeks for 6 cycles.
  EPOCH: EPOCH is given with Rituximab and bortezomib every 3 weeks for 6 cycles.
  Bortezomib (B): Bortezomib is given alone for one cycle. Bortezomib or observation: At the beginning of Part C, patients are randomized to receive bortezomib maintenance or be observed w/o bortezomib.
Arm/Group | All Participants
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.85 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time interval from start of treatment to documented evidence of disease progression. Progression is defined by at least one of the following: ≥50% increase in the sum of the products of at least two lymph nodes, appearance of new lymph nodes, ≥50% increase in the size of the liver and/or spleen as determined by measurement below the respective costal margin, appearance of new palpable hepatomegaly or splenomegaly that was not previously present, and ≥50% increase in the absolute number of circulating lymphocytes.The primary evaluation will be a Kaplan-Meier analysis with a two tailed log rank test.
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Bortezomib Maintenance: Bortezomib maintenance
  Bortezomib: Bortezomib is given with EPOCH and rituximab every 3 weeks for 6 cycles.
- Observation: Observation without bortezomib
- Not Randomized: Twenty-three patients were not randomized. Sixteen due to neuropathy and seven due to "other" reasons.
Arm/Group | Bortezomib Maintenance | Observation | Not Randomized
Number analyzed (Participants) | 14 | 16 | 23
Months | 27.2 [12.4 to 51.5] | 33.5 [20.3 to NA] — That is a statistical reason; since the OS was so high, the upper limit of confidence interval is undefined. | 7.8 [4.3 to 29.0]

2. Primary Outcome: Median Overall Survival (OS)
Description: Overall Survival is the time between the first day of treatment to the day of death. The primary evaluation will be a Kaplan-Meier analysis with a two tailed log rank test.
Time Frame: up to 9.9 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- EPOCH-R+Bortezomib: Combo chemo etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH)-Rituxan (R) + Bortezomib (B)
  Rituximab (R): Rituximab is given with etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) and bortezomib every 3 weeks for 6 cycles.
  EPOCH: EPOCH is given with Rituximab and bortezomib every 3 weeks for 6 cycles.
  Bortezomib (B): Bortezomib is given alone for one cycle.
Arm/Group | EPOCH-R+Bortezomib
Number analyzed (Participants) | 53
Months | 80.4 [66.6 to 89.0]

3. Primary Outcome: Overall Progression Free Survival
Description: Time interval from start of treatment to documented evidence of disease progression. Progression is defined by at least one of the following: ≥50% increase in the sum of the products of at least two lymph nodes, appearance of new lymph nodes, ≥50% increase in the size of the liver and/or spleen as determined by measurement below the respective costal margin, appearance of new palpable hepatomegaly or splenomegaly that was not previously present, and ≥50% increase in the absolute number of circulating lymphocytes.
Time Frame: up to 9.9 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EPOCH-R+Bortezomib
Number analyzed (Participants) | 53
Months | 29.3 [20.3 to 35.8]

4. Primary Outcome: Overall Survival
Description: as for outcome 2
Time Frame: up to 9.9 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bortezomib Maintenance | Observation | Not Randomized
Number analyzed (Participants) | 14 | 16 | 23
Months | 78.6 [47.2 to 92.5] | 87.5 [58.6 to 96.7] | 31.6 [4.9 to NA] — That is a statistical reason; since the OS was so high, the upper limit of confidence interval is undefined.

5. Secondary Outcome: Count of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 143 months and 7 days
Population: Participants are grouped together in one arm/group because most adverse events occurred during Part B, in which all participants received drug.
Measure: Count of Participants; unit: Participants
Arm/Group | EPOCH-R+Bortezomib
Number analyzed (Participants) | 53
Participants | 53

6. Secondary Outcome: Clinical Response
Description: Clinical response is assessed by the response criteria for lymphomas and is defined as a fraction of patients who have a complete response (CR) or a complete response (CR) + partial response (PR). A complete response is disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities (e.g. lactate dehydrogenase) definitely assignable to the lymphoma. Partial response is ≥50% decreased in the sum of the products of the greatest diameters of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Progressive disease is defined by at least one of the following: ≥50% increase in the sum of the products of at least two lymph nodes appearance of new lymph nodes, ≥50% increase in the size of the liver and/or spleen, ≥50% increase in the absolute number of circulating lymphocytes.
Time Frame: up to 22 weeks after initiation of therapy
Population: Participants are grouped together in one arm/group because this is the arm/group in which all participants received drug.
Measure: Number; unit: Percentage of patients
Arm/Group | EPOCH-R+Bortezomib
Number analyzed (Participants) | 53
Percentage of patients
  Overall Response (CR+PR) | 92.5
  Complete Response | 86.7
  Stable Disease | 3.8
  Progressive Disease | 1.9
  Not Evaluable | 1.9

ADVERSE EVENTS:
Time Frame: date treatment consent signed to date off study, approximately 143 months and 7 days
Description: Participants are grouped together in one arm/group because most adverse events occurred during Part B, in which all participants received drug.
Arm/Group | EPOCH-R+Bortezomib
All-Cause Mortality (participants affected / at risk) | 1/53
Serious Adverse Events (participants affected / at risk) | 21/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPOCH-R+Bortezomib (N=53)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 9 (11) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, CNS (Nervous system disorders) | 1 (1)
Hemorrhage, GI::Peritoneal cavity (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1)
Obstruction, GI::Colon (Gastrointestinal disorders) | 1 (1)
Obstruction, GI::Small bowel NOS (Gastrointestinal disorders) | 1 (2)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (2)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Perforation, GI::Colon (Gastrointestinal disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPOCH-R+Bortezomib (N=53)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 19 (39)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 16 (28)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 36 (92)
Alkaline phosphatase (Metabolism and nutrition disorders) | 16 (22)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 12 (18)
Anorexia (Metabolism and nutrition disorders) | 17 (21)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites (non-malignant) (Eye disorders) | 2 (2)
Ataxia (incoordination) (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 3 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 13 (23)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 2 (2)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4 (9)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 20 (69)
Cardiac General - Other (cardiac tamponade) (Cardiac disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 32 (50)
Constitutional Symptoms - Other (early satiety (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Creatinine (Metabolism and nutrition disorders) | 9 (15)
Cystitis (Renal and urinary disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Dermatology/Skin - Other (folliculitis) (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 30 (49)
Distension/bloating, abdominal (Gastrointestinal disorders) | 6 (7)
Dizziness (Nervous system disorders) | 21 (26)
Dry eye syndrome (Eye disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 5 (5)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 16 (22)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 27 (41)
Esophagitis (Gastrointestinal disorders) | 1 (1)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 35 (54)
Febrile neutropenia (fever of unknown origin (Infections and infestations) | 13 (15) — without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 14 (14)
Flatulence (Gastrointestinal disorders) | 3 (3)
Flu-like syndrome (General disorders) | 1 (1)
Gastrointestinal - Other (hiccups) (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 18 (48)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 6 (7)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 40 (48)
Heartburn/dyspepsia (Gastrointestinal disorders) | 9 (9)
Hemoglobin (Blood and lymphatic system disorders) | 53 (392)
Hemorrhage, GI::Anus (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI::Colon (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hemorrhage/Bleeding - Other vitreous hemorrhage) (Eye disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2 (9)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 15 (21)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Abdomen NOS
Infection (Infections and infestations) | 2 (4) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 1 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Colon
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Ileum
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (Infections and infestations) | 1 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Mucosa
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Oral cavity-gums (gingivitis)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Sinus
Infection (Infections and infestations) | 3 (3) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Skin (cellulitis)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Trachea
Infection - Other (sinusitis) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Abdomen NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Mucosa (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nerve-peripheral (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Oral cavity-gums (gingivitis) (Infections and infestations) | 3 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 4 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 2 (2)
Infection with unknown ANC::Soft tissue NOS (Infections and infestations) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 3 (3)
Insomnia (General disorders) | 18 (21)
Intra-operative injury::Muscle (Surgical and medical procedures) | 1 (1)
Laryngeal nerve dysfunction (Nervous system disorders) | 3 (5)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 53 (345)
Lymphopenia (Blood and lymphatic system disorders) | 53 (451)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 12 (22)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 13 (58)
Memory impairment (Nervous system disorders) | 1 (1)
Mood alteration::Agitation (Nervous system disorders) | 1 (1)
Mood alteration::Anxiety (Nervous system disorders) | 4 (4)
Mood alteration::Depression (Nervous system disorders) | 4 (4)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 23 (46)
Mucositis/stomatitis (clinical exam)::Stomach (Gastrointestinal disorders) | 3 (3)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 11 (12)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 4 (5)
Nail changes (Skin and subcutaneous tissue disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 27 (58)
Neurology - Other (autonomic neuropathy) (Nervous system disorders) | 3 (4)
Neuropathy: motor (Nervous system disorders) | 8 (9)
Neuropathy: sensory (Nervous system disorders) | 52 (93)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 53 (271)
Obstruction, GI::Ileum (Gastrointestinal disorders) | 1 (1)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 16 (27)
Pain - Other (Specify, Jaw-GCSF) (Nervous system disorders) | 8 (11)
Pain::Abdomen NOS (Gastrointestinal disorders) | 12 (14)
Pain::Back (Musculoskeletal and connective tissue disorders) | 11 (11)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 32 (61)
Pain::Cardiac/heart (Cardiac disorders) | 1 (1)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 7 (9)
Pain::Head/headache (Nervous system disorders) | 15 (20)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 10 (10)
Pain::Kidney (Renal and urinary disorders) | 1 (1)
Pain::Lymph node (Blood and lymphatic system disorders) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 9 (12)
Pain::Neuralgia/peripheral nerve (Nervous system disorders) | 12 (18)
Pain::Oral cavity (Gastrointestinal disorders) | 1 (1)
Pain::Pericardium (Cardiac disorders) | 1 (1)
Pain::Rectum (Gastrointestinal disorders) | 1 (1)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain::Urethra (Renal and urinary disorders) | 1 (2)
Palpitations (Cardiac disorders) | 3 (3)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 2 (2)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 13 (25)
Platelets (Blood and lymphatic system disorders) | 53 (419)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 (9)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 13 (24)
Proctitis (Gastrointestinal disorders) | 1 (1)
Prolapse of stoma, GI (Gastrointestinal disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (3)
Pulmonary/Upper Respiratory - Other (tachypnea) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16 (18)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Rigors/chills (General disorders) | 9 (11)
Seroma (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 7 (8)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 20 (44)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 2 (2)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 4 (6)
Supraventricular and nodal arrhythmia::Supraventricular arrhythmia NOS (Cardiac disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 5 (6)
Syncope (fainting) (Nervous system disorders) | 3 (3)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 13 (17)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 4 (4)
Thrombosis/thrombus/embolism (Vascular disorders) | 6 (8)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 7 (10)
Urinary frequency/urgency (Renal and urinary disorders) | 3 (3)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Ventricular arrhythmia::Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vessel injury-vein::Extremity-upper (Vascular disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Vision-photophobia (Eye disorders) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 12 (15)
Watery eye (epiphora, tearing) (Eye disorders) | 11 (14)
Weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 8 (13)
Gastrointestinal - Other (Stomatitis) (Gastrointestinal disorders) | 2 (3)
Gastrointestinal - Other (Stomatitis - Ulcer on tongue) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Thrush) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Stomatitis/pharyngitis) (Gastrointestinal disorders) | 1 (1)
Neurology - Other (fall) (Nervous system disorders) | 1 (1)
Pain - Other (neuropathic) (Nervous system disorders) | 1 (1)
Pain - Other (pain Lt biopsy site) (General disorders) | 1 (1)
Pain - Other (pain R arm) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other (pain in extremity) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other (skin/shingles) (Skin and subcutaneous tissue disorders) | 1 (1)
Pain - Other (sore throat) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain - Other (surgical site) (Surgical and medical procedures) | 1 (1)
Pain - Other (arm) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other (extremities) (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT00114738/Prot_SAP_002.pdf
  • Informed Consent Form: Standard Consent (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT00114738/ICF_003.pdf